CLINICAL TRIAL: NCT02885298
Title: Prospective Observational Study of the Effect of Upright Patient Positioning on Intubation Success Rates at Two Academic Emergency Departments
Brief Title: Effect of Upright Patient Positioning on Intubation Success
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Joseph Turner, Assistant Professor of Clinical Emergency Medicine, Indiana University
Other Study IDs: 1405954059
Record Dates: First submitted 2016-08-24; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Supine intubations (0-10 degrees): Intubations performed with patient positioned 0-10 degrees. Patient supine.
  Interventions: Procedure: Upright intubation
- Inclined (11-44 degrees): Intubations performed with 11-44 degrees of elevation.
  Interventions: Procedure: Upright intubation
- Upright (45 degrees or greater): intubations performed with patient elevated to 45 degrees or greater
  Interventions: Procedure: Upright intubation

INTERVENTIONS:
Procedure: Upright intubation — Upright Intubation procedure performed with patient elevated above the supine position. Defined as upright greater to or equal to 45 degrees or inclined 10-44 degrees

SUMMARY:
Endotracheal intubation is most commonly taught and performed with the patient supine. Recent literature suggests that elevating the patient's head to a more upright position may decrease peri-intubation complications. However, there is little data on success rates of upright intubation in the emergency department. The goal of this study was to measure the association of head positioning with intubation success rates among emergency medicine residents.

DETAILED DESCRIPTION:
Endotracheal intubation is most commonly taught and performed with the patient supine. Recent literature suggests that elevating the patient's head to a more upright position may decrease peri-intubation complications. However, there is little data on success rates of upright intubation in the emergency department. The goal of this study was to measure the association of head positioning with intubation success rates among emergency medicine residents. Study design was a prospective observational study. Residents performing intubation recorded the angle of the head of the bed, and the number of attempts required for successful intubation was recorded by faculty and respiratory therapists. The primary outcome of first past success was calculated with respect to three groups: 0-10 degrees (supine), 11-44 degrees (inclined), and ≥45 degrees (upright); first past success was also analyzed in 5 degree angle increments.

ELIGIBILITY:
Inclusion Criteria:

* Adult medical intubations in which the intubating resident and supervising faculty both consented to study participation.

Exclusion Criteria:

* Pediatric patients
* Obstetric patients
* Trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubation events that were eligible for enrollment included adult medical intubations performed at participating hospitals in which the intubating resident and supervising faculty both consented to study participation.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
First Pass Success | Immediately at the time of the procedure
  An attempt was defined as anytime the laryngoscope blade was placed in the patient's mouth. At the beginning of the study residents, faculty, and RTs were educated on this definition.

SECONDARY OUTCOMES:
overall success rate of orotracheal intubation overall success rate of orotracheal intubation overall success rate of intubation | Immediately at the time of the procedure
  endotracheal tube in place
Time required for successful intubation | Immediately at the time of the procedure
  endotracheal tube in place
esophageal intubation | Immediately at the time of the procedure
  endotracheal tube determined to be positioned in esophagus rather
cardiac arrest within 30 minutes of the intubation attempt | cardiac arrest within 30 minutes of intubation
decrease in oxygen saturation during the procedure | Immediately at the time of the procedure
best Cormack-Lehane view | Immediately at the time of the procedure
  Cormack-Lehane view is a scale that is used to describe the amount of vocal cords visualized during the procedure
best Percent of Glottic Opening (POGO) | obtained during the procedure
  Percent of glottis opening refers to the percentage of vocal cords and surrounding anatomy which can be seen during the procedure
Resident Satisfaction with Positioning | following procedure
  survey completed following the procedure by provider regarding satisfaction
death in ED | While in the emergency department (1 hour up to 1 day)
death within 5 days of intubation | Death within 5 days following intubation
  any cause of death within 5 days after intubation
New pneumonia | within 5 days following intubation
  new pneumonia developed within 5 days following an intubation. Not present on admission.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Turner, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szmuk P, Ezri T, Evron S, Roth Y, Katz J. A brief history of tracheostomy and tracheal intubation, from the Bronze Age to the Space Age. Intensive Care Med. 2008 Feb;34(2):222-8. doi: 10.1007/s00134-007-0931-5. Epub 2007 Nov 13. PMID 17999050
- [Background] Mouton WG, Bessell JR, Maddern GJ. Looking back to the advent of modern endoscopy: 150th birthday of Maximilian Nitze. World J Surg. 1998 Dec;22(12):1256-8. doi: 10.1007/s002689900555. PMID 9841754
- [Background] Burkle CM, Zepeda FA, Bacon DR, Rose SH. A historical perspective on use of the laryngoscope as a tool in anesthesiology. Anesthesiology. 2004 Apr;100(4):1003-6. doi: 10.1097/00000542-200404000-00034. No abstract available. PMID 15087639
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Jaber S, Amraoui J, Lefrant JY, Arich C, Cohendy R, Landreau L, Calvet Y, Capdevila X, Mahamat A, Eledjam JJ. Clinical practice and risk factors for immediate complications of endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Crit Care Med. 2006 Sep;34(9):2355-61. doi: 10.1097/01.CCM.0000233879.58720.87. PMID 16850003
- [Background] Li J, Murphy-Lavoie H, Bugas C, Martinez J, Preston C. Complications of emergency intubation with and without paralysis. Am J Emerg Med. 1999 Mar;17(2):141-3. doi: 10.1016/s0735-6757(99)90046-3. PMID 10102312
- [Background] Schwartz DE, Matthay MA, Cohen NH. Death and other complications of emergency airway management in critically ill adults. A prospective investigation of 297 tracheal intubations. Anesthesiology. 1995 Feb;82(2):367-76. doi: 10.1097/00000542-199502000-00007. PMID 7856895
- [Background] Mort TC. Complications of emergency tracheal intubation: hemodynamic alterations--part I. J Intensive Care Med. 2007 May-Jun;22(3):157-65. doi: 10.1177/0885066607299525. PMID 17562739
- [Background] Mort TC. Complications of emergency tracheal intubation: immediate airway-related consequences: part II. J Intensive Care Med. 2007 Jul-Aug;22(4):208-15. doi: 10.1177/0885066607301359. PMID 17712056
- [Background] Griesdale DE, Bosma TL, Kurth T, Isac G, Chittock DR. Complications of endotracheal intubation in the critically ill. Intensive Care Med. 2008 Oct;34(10):1835-42. doi: 10.1007/s00134-008-1205-6. Epub 2008 Jul 5. PMID 18604519
- [Background] Dargin JM, Emlet LL, Guyette FX. The effect of body mass index on intubation success rates and complications during emergency airway management. Intern Emerg Med. 2013 Feb;8(1):75-82. doi: 10.1007/s11739-012-0874-x. Epub 2012 Nov 25. PMID 23184440
- [Background] Jaber S, Jung B, Corne P, Sebbane M, Muller L, Chanques G, Verzilli D, Jonquet O, Eledjam JJ, Lefrant JY. An intervention to decrease complications related to endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Intensive Care Med. 2010 Feb;36(2):248-55. doi: 10.1007/s00134-009-1717-8. Epub 2009 Nov 17. PMID 19921148
- [Background] Kim GW, Koh Y, Lim CM, Han M, An J, Hong SB. Does medical emergency team intervention reduce the prevalence of emergency endotracheal intubation complications? Yonsei Med J. 2014 Jan;55(1):92-8. doi: 10.3349/ymj.2014.55.1.92. PMID 24339292
- [Background] Khandelwal N, Khorsand S, Mitchell SH, Joffe AM. Head-Elevated Patient Positioning Decreases Complications of Emergent Tracheal Intubation in the Ward and Intensive Care Unit. Anesth Analg. 2016 Apr;122(4):1101-7. doi: 10.1213/ANE.0000000000001184. PMID 26866753
- [Background] Lane S, Saunders D, Schofield A, Padmanabhan R, Hildreth A, Laws D. A prospective, randomised controlled trial comparing the efficacy of pre-oxygenation in the 20 degrees head-up vs supine position. Anaesthesia. 2005 Nov;60(11):1064-7. doi: 10.1111/j.1365-2044.2005.04374.x. PMID 16229689
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Ramkumar V, Umesh G, Philip FA. Preoxygenation with 20 masculine head-up tilt provides longer duration of non-hypoxic apnea than conventional preoxygenation in non-obese healthy adults. J Anesth. 2011 Apr;25(2):189-94. doi: 10.1007/s00540-011-1098-3. Epub 2011 Feb 4. PMID 21293885
- [Background] Lee BJ, Kang JM, Kim DO. Laryngeal exposure during laryngoscopy is better in the 25 degrees back-up position than in the supine position. Br J Anaesth. 2007 Oct;99(4):581-6. doi: 10.1093/bja/aem095. Epub 2007 Jul 4. PMID 17611252
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Diggs LA, Viswakula SD, Sheth-Chandra M, De Leo G. A pilot model for predicting the success of prehospital endotracheal intubation. Am J Emerg Med. 2015 Feb;33(2):202-8. doi: 10.1016/j.ajem.2014.11.020. Epub 2014 Nov 20. PMID 25488339
- [Background] Neligan PJ, Porter S, Max B, Malhotra G, Greenblatt EP, Ochroch EA. Obstructive sleep apnea is not a risk factor for difficult intubation in morbidly obese patients. Anesth Analg. 2009 Oct;109(4):1182-6. doi: 10.1213/ane.0b013e3181b12a0c. PMID 19762747
- [Background] Tremblay MH, Williams S, Robitaille A, Drolet P. Poor visualization during direct laryngoscopy and high upper lip bite test score are predictors of difficult intubation with the GlideScope videolaryngoscope. Anesth Analg. 2008 May;106(5):1495-500, table of contents. doi: 10.1213/ane.0b013e318168b38f. PMID 18420866
- Available data/document: Study Protocol — https://drive.google.com/drive/folders/0B5w-TjIZHObhSWxqbElCUmxINnc — Study protocol can be provided via email if requested. Please email turnjose@iu.edu